CLINICAL TRIAL: NCT01707550
Title: Observational, Non-interventional Survey of Renal Allograft Recipients Receiving CellCept as Part of Their Immunosuppressive Protocol
Brief Title: An Observational Study of CellCept (Mycophenolate Mofetil) in Renal Allograft Recipients
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25048
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational survey study will capture all renal transplant patients in Serbia who are currently receiving CellCept (mycophenolate mofetil) as part of their immunosuppressive protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Recipients of renal allograft
* Patients receiving CellCept

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal allograft recipients receiving CellCept as part of their immunosuppressive protocol
Sampling Method: Probability Sample
Enrollment: 414 (Actual)
Dates: Start 2009-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Average dose of CellCept used in immunosuppressive protocols in Serbia | 9 months
Average dose of concomitant immunosuppressive drugs | 9 months

SECONDARY OUTCOMES:
Average duration of post-transplant period for patients in Serbia receiving CellCept | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Serbia (3):
  - Belgrade
  - Niš
  - Novi Sad